CLINICAL TRIAL: NCT01270984
Title: Open Label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetic Characteristics of Luckyvec 400mg Tablet, in Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetic Characteristics of Luckyvec 400mg Tablet, in Healthy Subjects
Acronym: Imatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 131HPS10D
Record Dates: First submitted 2011-01-04; First posted 2011-01-06 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Myeloid Leukemia; Gastrointestinal Stromal Tumors
Keywords: Imatinib mesylate; Pharmacokinetics; Healthy volunteers
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Luckyvec 400mg film coated tablet (Experimental): 400mg/tablet, PO, 1 tablet once daily for Period I & II D1(crossover)
  Interventions: Drug: Luckyvec 400mg film coated tablet
- Glivec 100mg film coated tablet (Active Comparator): 100mg/tablet, PO, 4 tablets once daily for Period I & II D1(crossover)
  Interventions: Drug: Glivec 100mg film coated tablet

INTERVENTIONS:
Drug: Luckyvec 400mg film coated tablet — •400mg/tablet, PO, 1 tablet once daily for Period I & II D1(crossover)
  Other Names: Luckyvec
  Arms: Luckyvec 400mg film coated tablet
Drug: Glivec 100mg film coated tablet — •100mg/tablet, PO, 4 tablets once daily for Period I & II D1(crossover)
  Other Names: Glivec
  Arms: Glivec 100mg film coated tablet

SUMMARY:
The purpose of this study is to evaluate safety and tolerance by comparing pharmacokinetic characteristics between the Luckyvec 400mg tablet(x 1T) and Glivec 100mg(x 4T) when administered a single-dose to healthy volunteers.

DETAILED DESCRIPTION:
Healthy volunteers are administrated single-dose over the period I and II (Crossover) of Luckyvec 400mg tablet(x 1T) and Glivec 100mg(x 4T)as of Imatinib 400mg.

Every time before and after each medication, PK parameters and safety of Luckyvec 400mg tablet and Glivec 100mg is performed using a blood sample and conducting some tests(Laboratory test, V/S, Physical Examination, etc) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 aged and 45 aged in healthy males
* BMI: 18~29.9 kg/m2, (BMI = (체중 [kg])/(height [m])2)
* Agreement with written informed consent

Exclusion Criteria:

* Clinically significant cardiovascular system, pulmonary system, liver system, renal system, blood system, gastrointestinal system, immune system, skin system, nervous system or mental disease(Past history or present)
* Subject with symptoms of acute disease within 28 days of starting administration of investigational drug
* Subject with known for history which affect on the ADME of drug
* Clinically significant active chronic disease
* Inadequate result of laboratory test

  * AST/ALT > 1.5 x UNL
  * Total bilirubin > 1.5 x UNL
* Positive reaction in the HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL test
* Taking ETC(ethical the counter)medicine within 14 days
* Taking OTC(Over the counter)medicine including oriental medicine within 7 days
* Clinically significant allergic disease(Except for mild allergic rhinitis and dermatits seems to be not need for medication)
* Subject with known for hypersensitivity reaction to imatinib analog
* Not able to taking the institutional standard meal
* Previously make whole blood donation within 60 days or component blood donation within 20 days
* Previously have blood transfusion within 30 days
* Previously participated in other trial within 30 days
* Continued to be taking caffeine (caffeine > 5 cup/day), drinking(alcohol > 30 g/day) and severe heavy smoker (cigarette > 1/2 pack per day)
* An impossible one who participates in clinical trial by investigator's decision including for reason of laboratory test result

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of Luckyvec 400mg tablet and Glivec 100mg tablet in healthy subjects | 0-72hr

SECONDARY OUTCOMES:
To evaluate the safety of Luckyvec 400mg tablet and Glivec 100mg tablet from vital signs, physical exam, ECG, laboratory test, adverse event and so on. | 0-72hr

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, Principal Investigator — jypark21@korea.ac.kr
Locations (1):
- The Korea University Anam Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim KA, Park SJ, Kim C, Park JY. Single-dose, randomized crossover comparisons of different-strength imatinib mesylate formulations in healthy Korean male subjects. Clin Ther. 2013 Oct;35(10):1595-602. doi: 10.1016/j.clinthera.2013.08.008. Epub 2013 Sep 21. PMID 24060561